CLINICAL TRIAL: NCT05469451
Title: Effect of Diode Laser (940nm) on Total Relief of Dental Crowding and Pain Perception in Orthodontics: Randomized Clinical Trial (RCT)
Brief Title: Effect of the Diode Laser (940nm) on Orthodontics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Universitaria CIEO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UniCIEOLaser01
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Low Level Laser Therapy; Pain; Crowding, Tooth
Keywords: Low-Level Light Therapy; Malocclusion; Orthodontics; Pain
MeSH Terms: conditions — Pain; Malocclusion | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: 50 randomized subjects, 25 per group, seen during the alignment phase with ages between 20 and 40 years, male or female, with all lower permanent teeth or at least 36 to 46, with Little's irregularity index 3mm to 6mm, without prior orthodontic treatment, periodontally stable, non-smokers and who voluntarily agreed to participate in the study by signing the informed consent.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patients participating in the clinical trial, the statistician, the students and the study operators who are going to measure Little's irregularity index will be blinded to the interventions, except the principal investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: irradiated with low power laser (940nm) (Experimental): Irradiated with a low power density laser of 940 (nm), 100 megawatt, which will be calibrated and the result of the calibration will be checked with the use of the power meter. The equipment used will be a diode laser (BIOLASE™), the area to be irradiated will be the anterior segment of the lower arch, each tooth will be irradiated for a time of 10 seconds on the vestibular surfaces of the teeth and 10 seconds on the lingual surfaces of the teeth, both at gingival level and at apical level in scanning mode.
  Interventions: Procedure: Low level laser therapy
- Group 2: Simulated that they were irradiated. (Placebo Comparator): Group 2: it was simulated that they were irradiated.
  Interventions: Procedure: Low level laser therapy

INTERVENTIONS:
Procedure: Low level laser therapy — Irradiated with a low power density laser of 940 (nm), 100 megawatt, which will be calibrated and the result of the calibration will be checked with the use of the power meter. The equipment used will be a diode laser (BIOLASE™), the area to be irradiated will be the anterior segment of the lower arch, each tooth will be irradiated for a time of 10 seconds on the vestibular surfaces of the teeth and 10 seconds on the lingual surfaces of the teeth, both at gingival level and at apical level in scanning mode.

SUMMARY:
To evaluate the effect of the low power density 940nm diode laser in the total relief of dental crowding during the alignment phase and the perception of pain in patients who initiate orthodontic treatment.

DETAILED DESCRIPTION:
Objectives: To evaluate the effect of the low power density 940nm diode laser in the total relief of dental crowding during the alignment phase and the perception of pain in patients who initiate orthodontic treatment.

Design: Randomized clinical trial. Setting: orthodontic treatment from the Orthodontic postgraduate course at the CIEO University (CIEO), located in the city of Bogotá, Colombia Participants: 50 randomized subjects, 25 per group, seen during the alignment phase with ages between 20 and 40 years, male or female, with all lower permanent teeth or at least 36 to 46, with Little's irregularity index 3mm to 6mm, without prior orthodontic treatment, periodontally stable, non-smokers and who voluntarily agreed to participate in the study by signing the informed consent. Patients with a history of long-term medications that interfere with bone metabolism and / or pain synthesis (bisphosphonates, anti-inflammatory or analgesic drugs and hormonal supplements, with systemic diseases (Diabetes, hyperthyroidism, disease with bone metabolism) were excluded. , pregnant women, infants and patients who, during the alignment phase, require the implementation of metal ligatures, springs to expand spaces and lace back uses in the technique.

Intervention: group 1 irradiated with low power laser (940nm) and. Group 2: it was simulated that they were irradiated. The therapeutic laser was applied for a time of 10 seconds on the buccal surfaces of the teeth and 10 seconds on the lingual surfaces of the teeth, both at the gingival level and at the apical level in scanning mode, on the day of cementation of the appliance and subsequently every fifteen days for 3 months.

Main outcome measures: total relief of dental crowding measured through the little index in digital models and pain perception through the visual analog scale.

Randomization: Four patients were randomized with the randomized blocks technique.

Blinding (masking): The patients participating in the clinical trial, the statistician, the students and the study operators who are going to measure Little's irregularity index will be blinded to the interventions, except the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 20 and 40 years
* Male or female
* All lower permanent teeth or at least 36 to 46
* Little's irregularity index 3mm to 6mm
* Without prior orthodontic treatment
* Periodontally stable
* Non-smokers
* Voluntarily agreed to participate in the study by signing the informed consent

Exclusion Criteria:

* Patients with a history of long-term medications that interfere with bone metabolism and / or pain synthesis (bisphosphonates, anti-inflammatory or analgesic drugs and hormonal supplements
* Systemic diseases (Diabetes, hyperthyroidism, disease with bone metabolism)
* Pregnant women
* Infants
* Patients who, during the alignment phase, require the implementation of metal ligatures, springs to expand spaces and lace back uses in the technique.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-20 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Total relief of dental crowding | 3 months
  This was measured as the resolution of anterior crowding in the lower arch calculated by the difference of Little's irregularity index, the distance in millimeters between the contact points from mesial of the canine to mesial of the contralateral canine in the lower arch in the digitized models in each of the established times. Perfect alignment from the mesial aspect of the left canine to the mesial aspect of the right canine would theoretically have a score of 0, with greater crowding represented by greater displacement and thus a higher index score.

SECONDARY OUTCOMES:
Pain perception | 3 months
  by means of the visual analog scale that represents the intensity of the pain in a line from 0 to 10. At one end there is the phrase "no pain" and at the opposite end "the worst pain imaginable". A value of less than 4 on the VAS means mild or mild-moderate pain, a value between 4 and 6 implies the presence of moderate-severe pain, and a value greater than 6 implies the presence of very intense pain.

CONTACTS AND LOCATIONS:
Overall Officials: Diana M Montoya, MSc, Study Chair — Fundación Universitaria CIEO
Locations (1):
- Fundación Universitaria UniCIEO, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gounder R, Gounder S. Laser Science and its Applications in Prosthetic Rehabilitation. J Lasers Med Sci. 2016 Fall;7(4):209-213. doi: 10.15171/jlms.2016.37. Epub 2016 Oct 27. PMID 28491254
- [Background] Demirsoy KK, Kurt G. Use of Laser Systems in Orthodontics. Turk J Orthod. 2020 May 22;33(2):133-140. doi: 10.5152/TurkJOrthod.2020.18099. eCollection 2020 Jun. PMID 32637195
- [Background] Chen H, Han B, Jiang R, Su H, Feng T, Teng F, Xu T. PASS versus MBT for evaluation of anchorage control in three-dimensional measurements: a randomized controlled trial. Eur J Orthod. 2021 Jan 29;43(1):113-119. doi: 10.1093/ejo/cjaa021. PMID 32255178
- [Background] Scott P, Sherriff M, Dibiase AT, Cobourne MT. Perception of discomfort during initial orthodontic tooth alignment using a self-ligating or conventional bracket system: a randomized clinical trial. Eur J Orthod. 2008 Jun;30(3):227-32. doi: 10.1093/ejo/cjm131. Epub 2008 Mar 13. PMID 18339656
- [Background] Little RM. The irregularity index: a quantitative score of mandibular anterior alignment. Am J Orthod. 1975 Nov;68(5):554-63. doi: 10.1016/0002-9416(75)90086-x. PMID 1059332
- [Background] MOORREES CF, REED RB. Biometrics of crowding and spacing of the teeth in the mandible. Am J Phys Anthropol. 1954 Mar;12(1):77-88. doi: 10.1002/ajpa.1330120120. No abstract available. PMID 13148326
- [Background] Shaughnessy T, Kantarci A, Kau CH, Skrenes D, Skrenes S, Ma D. Intraoral photobiomodulation-induced orthodontic tooth alignment: a preliminary study. BMC Oral Health. 2016 Jan 13;16:3. doi: 10.1186/s12903-015-0159-7. PMID 26762247
- [Background] Proffit WR, Ackerman JL. Rating the characteristics of malocclusion: a systematic approach for planning treatment. Am J Orthod. 1973 Sep;64(3):258-69. doi: 10.1016/0002-9416(73)90019-5. No abstract available. PMID 4579697
- [Background] Camacho AD, Velasquez Cujar SA. Dental movement acceleration: Literature review by an alternative scientific evidence method. World J Methodol. 2014 Sep 26;4(3):151-62. doi: 10.5662/wjm.v4.i3.151. eCollection 2014 Sep 26. PMID 25332914
- [Background] Peck H, Peck S. An index for assessing tooth shape deviations as applied to the mandibular incisors. Am J Orthod. 1972 Apr;61(4):384-401. doi: 10.1016/0002-9416(72)90302-8. No abstract available. PMID 4501985
- [Background] Li B, Zhao ZH. [Adjunctive interventions to accelerate orthodontic tooth movement]. Hua Xi Kou Qiang Yi Xue Za Zhi. 2019 Dec 1;37(6):648-655. doi: 10.7518/hxkq.2019.06.014. Chinese. PMID 31875445
- [Background] Diddige R, Negi G, Kiran KVS, Chitra P. Comparison of pain levels in patients treated with 3 different orthodontic appliances - a randomized trial. Med Pharm Rep. 2020 Jan;93(1):81-88. doi: 10.15386/mpr-1311. Epub 2020 Jan 31. PMID 32133451
- [Background] Asiry MA. Biological aspects of orthodontic tooth movement: A review of literature. Saudi J Biol Sci. 2018 Sep;25(6):1027-1032. doi: 10.1016/j.sjbs.2018.03.008. Epub 2018 Mar 14. PMID 30174498
- [Background] Fernandes LM, Ogaard B, Skoglund L. Pain and discomfort experienced after placement of a conventional or a superelastic NiTi aligning archwire. A randomized clinical trial. J Orofac Orthop. 1998;59(6):331-9. doi: 10.1007/BF01299769. English, German. PMID 9857602
- [Background] Long H, Wang Y, Jian F, Liao LN, Yang X, Lai WL. Current advances in orthodontic pain. Int J Oral Sci. 2016 Jun 30;8(2):67-75. doi: 10.1038/ijos.2016.24. PMID 27341389
- [Background] Fleming PS, Dibiase AT, Sarri G, Lee RT. Pain experience during initial alignment with a self-ligating and a conventional fixed orthodontic appliance system. A randomized controlled clinical trial. Angle Orthod. 2009 Jan;79(1):46-50. doi: 10.2319/121007-579.1. PMID 19123718
- [Background] Yassaei S, Aghili H, Afshari JT, Bagherpour A, Eslami F. Effects of diode laser (980 nm) on orthodontic tooth movement and interleukin 6 levels in gingival crevicular fluid in female subjects. Lasers Med Sci. 2016 Dec;31(9):1751-1759. doi: 10.1007/s10103-016-2045-1. Epub 2016 Sep 28. PMID 27680969
- [Background] Jahanbin A, Hasanzadeh N, Khaki S, Shafaee H. Comparison of self-ligating Damon3 and conventional MBT brackets regarding alignment efficiency and pain experience: A randomized clinical trial. J Dent Res Dent Clin Dent Prospects. 2019 Fall;13(4):281-288. doi: 10.15171/joddd.2019.043. PMID 32190212
- [Background] Sonesson M, De Geer E, Subraian J, Petren S. Efficacy of low-level laser therapy in accelerating tooth movement, preventing relapse and managing acute pain during orthodontic treatment in humans: a systematic review. BMC Oral Health. 2016 Jul 7;17(1):11. doi: 10.1186/s12903-016-0242-8. PMID 27431504
- [Background] El-Angbawi A, McIntyre GT, Fleming PS, Bearn DR. Non-surgical adjunctive interventions for accelerating tooth movement in patients undergoing fixed orthodontic treatment. Cochrane Database Syst Rev. 2015 Nov 18;2015(11):CD010887. doi: 10.1002/14651858.CD010887.pub2. PMID 26576758
- [Background] Isola G, Matarese M, Briguglio F, Grassia V, Picciolo G, Fiorillo L, Matarese G. Effectiveness of Low-Level Laser Therapy during Tooth Movement: A Randomized Clinical Trial. Materials (Basel). 2019 Jul 8;12(13):2187. doi: 10.3390/ma12132187. PMID 31288379
- [Background] Ureturk SE, Sarac M, Firatli S, Can SB, Guven Y, Firatli E. The effect of low-level laser therapy on tooth movement during canine distalization. Lasers Med Sci. 2017 May;32(4):757-764. doi: 10.1007/s10103-017-2159-0. Epub 2017 Mar 14. PMID 28289894
- [Background] Elkattan AE, Gheith M, Fayed MS, Yazeed MAE, Farrag AH, Khalil WKB. Effects of Different Parameters of Diode Laser on Acceleration of Orthodontic Tooth Movement and Its Effect on Relapse: An Experimental Animal Study. Open Access Maced J Med Sci. 2019 Feb 10;7(3):412-420. doi: 10.3889/oamjms.2019.089. eCollection 2019 Feb 15. PMID 30834013
- [Background] AlSayed Hasan MMA, Sultan K, Hamadah O. Low-level laser therapy effectiveness in accelerating orthodontic tooth movement: A randomized controlled clinical trial. Angle Orthod. 2017 Jul;87(4):499-504. doi: 10.2319/062716-503.1. Epub 2016 Nov 21. PMID 27869476
- [Background] Varella AM, Revankar AV, Patil AK. Low-level laser therapy increases interleukin-1beta in gingival crevicular fluid and enhances the rate of orthodontic tooth movement. Am J Orthod Dentofacial Orthop. 2018 Oct;154(4):535-544.e5. doi: 10.1016/j.ajodo.2018.01.012. PMID 30268264
- [Background] Al-Jundi A, Sakka S, Riba H, Ward T, Hanna R. Efficiency of Er:YAG utilization in accelerating deep bite orthodontic treatment. Laser Ther. 2018 Sep 30;27(3):193-202. doi: 10.5978/islsm.27_18-OR-15. PMID 32158065
- [Background] Qamruddin I, Alam MK, Mahroof V, Fida M, Khamis MF, Husein A. Effects of low-level laser irradiation on the rate of orthodontic tooth movement and associated pain with self-ligating brackets. Am J Orthod Dentofacial Orthop. 2017 Nov;152(5):622-630. doi: 10.1016/j.ajodo.2017.03.023. PMID 29103440
- [Background] Miles P. Accelerated orthodontic treatment - what's the evidence? Aust Dent J. 2017 Mar;62 Suppl 1:63-70. doi: 10.1111/adj.12477. PMID 28297096